CLINICAL TRIAL: NCT02838498
Title: Practice With ERCP Mechanical Simulator (EMS) Improves Basic ERCP Skills of Novice Surgical Trainees
Brief Title: Practice With Simulator Improves Basic ERCP Skills of Surgical Trainees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hepatopancreatobiliary Surgery Institute of Gansu Province (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Surgical ERCP EMS training
Record Dates: First submitted 2016-07-17; First posted 2016-07-20 (Estimated); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Hands-on Training
Keywords: ERCP; EMS; Cannulation; Successful rate; Trainee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive EMS training group (Experimental): Device: ERCP mechanical simulator training EMS group was coached (by JWL) on how to use the EMS, and then practiced with supervision by a senior surgeon biliary endoscopist (WBM). Trainees practiced for a total of 20 hours performing basic maneuvers including scope insertion 2 hours, scope positioning 6 hours, selective guide wire cannulation of common bile duct (CBD) stricture or pancreatic duct (PD) 10 hours and placement of a biliary stent 2 hours.
  All trainees received hands-on supervised clinical ERCP practice on patients. Time taken to perform ERCP procedures was documented. Trainees received verbal instructions, hands-on assistance from the trainer in performing the clinical procedure. If the trainee still failed after 20 minutes, the trainer took over.
  Interventions: Device: ERCP Mechanical Simulator (EMS)
- Routine ERCP training group (No Intervention): Other: Routine ERCP training group All trainees received hands-on supervised clinical ERCP practice on patients. Time taken to perform ERCP procedures was documented. Trainees received verbal instructions, hands-on assistance from the trainer in performing the clinical procedure. If the trainee still failed after 20 minutes, the trainer took over.

INTERVENTIONS:
Device: ERCP Mechanical Simulator (EMS) — Hands on EMS training
  Arms: Intensive EMS training group

SUMMARY:
To test the benefits of ERCP Mechanical Simulator (EMS) practice in improving ERCP cannulation success rate of novice surgical trainees.

DETAILED DESCRIPTION:
Practicing Endoscopic Retrograde Cholangiopancreatography (ERCP) procedures using the EMS provides opportunities for novice endoscopists to learn basic ERCP skills without a patient. In two randomized controlled trials (RCT), coached EMS practice increased selective bile duct cannulation success rate of novice endoscopists. Surgical trainees do not have sufficient endoscopy experience to meet the perceived basic requirement for ERCP training. However, ERCP is done with a side-viewing scope and even experienced GI trainees have difficult initially mastering the basic skill with scope manipulation and cannulation. It is not known whether EMS can provide additional benefit to novice surgical ERCP trainees.

ELIGIBILITY:
Inclusion Criteria:

* No experienced surgical trainees receiving ERCP training

Exclusion Criteria:

* Experienced surgical ERCP trainees or who are not receiving ERCP training

Min Age: 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-07; Primary Completion 2018-12-26 (Actual); Study Completion 2018-12-26 (Actual)

PRIMARY OUTCOMES:
Success rate of bile duct cannulation | 12 months
  Trainees received verbal instructions, hands-on assistance from the trainer no more than three times in performing the clinical procedure. The trainer took over if the trainee still failed after 20 minutes.

SECONDARY OUTCOMES:
Intubation time before cannulation | 12 months
  during the scope explored to cannulation
Successful cannulation time from first achieve the papilla | 12 months
  the time between the first achieve the papilla to cannulate successfully
Total time | 12 months
  From scope explored to withdraw
performance score of selective cannulation | 12 months
  The ability of trainees to perform solo diagnostic biliary cannulation and deep cannulation
Complication rate | 12 months
  The rate of major complications
Trainer assessment | 12 months
  Subjective competency graded by supervising physicians as above average, average or below average based on objective criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Xun Li, M.D., Ph. D., Principal Investigator — Hepatopancreatobiliary Surgery Institute of Gansu Province
Locations (1):
- Hepatopancreatobiliary Surgery Institute of Gansu Province, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Liao WC, Leung JW, Wang HP, Chang WH, Chu CH, Lin JT, Wilson RE, Lim BS, Leung FW. Coached practice using ERCP mechanical simulator improves trainees' ERCP performance: a randomized controlled trial. Endoscopy. 2013 Oct;45(10):799-805. doi: 10.1055/s-0033-1344224. Epub 2013 Jul 29. PMID 23897401
- [Result] Lim BS, Leung JW, Lee J, Yen D, Beckett L, Tancredi D, Leung FW. Effect of ERCP mechanical simulator (EMS) practice on trainees' ERCP performance in the early learning period: US multicenter randomized controlled trial. Am J Gastroenterol. 2011 Feb;106(2):300-6. doi: 10.1038/ajg.2010.411. Epub 2010 Oct 26. PMID 20978485